CLINICAL TRIAL: NCT01048463
Title: Phase 3 Study of Enteral Nutrition Rich in Eicosapentaenoic Acid in Patients Receiving Chemotherapy for Gastric Cancer or Colorectal Cancer
Brief Title: Effect of Enteral Nutrition Rich in Eicosapentaenoic Acid (EPA) on Patients Receiving Chemotherapy for GI Tumor
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Guanqing Sun, Dr., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPACT
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Gastric Cancer; Colorectal Cancer; Chemotherapy
Keywords: gastric cancer; colorectal cancer; chemotherapy; eicosapentaenoic acid; enteral nutrition
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms | interventions — Eicosapentaenoic Acid; Gelatin; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EN (Placebo Comparator): The subjects take in 150g of Nutriall per day. Oral administration of the liquid is divided into 3 times per day. The treatment lasts for 21d. During the test period patients are treated with the first course of XELOX.
  Interventions: Drug: Nutriall; Drug: Placebo; Drug: Chemotherapy
- ENLDEPA (Experimental): The subjects take in the same dose of Nutriall for the same duration as those in EN group. In addition, they take in 3 grams of EPA per day during the 21 days of treatment. The patients are treated with the first course of XELOX.
  Interventions: Drug: Nutriall; Drug: LDEPA; Drug: Chemotherapy
- ENHDPEA (Experimental): The subjects take in the same dose of supportan for the same duration as those in EN group. In addition, they take in 6 grams of EPA per day during the 21 days of treatment. The patients are treated with the first course of XELOX.
  Interventions: Drug: Nutriall; Drug: HDEPA; Drug: Chemotherapy

INTERVENTIONS:
Drug: Nutriall — The subjects take in 150g of Nutriall (Produced by Guangdong Academy of Agriculture Science. Every 50 grams of nutriall contains 9.3mg of VitC and 0.8mg of VitE) per day. Oral administration of the liquid is divided into 3 times per day. The treatment lasts for 21d.
  Other Names: Complete Enteral Nutrition Emulsion for cancer patients
Drug: LDEPA — The subjects take in 24 pils of EPA capsule per day. The medium is gelatine. Each capsule contains 0.125g of EPA and 0.125g of olive oil. The capsules are provided by nutritional department of our institute). The treatment lasts for 21d.
  Other Names: Eicosapentaenoic acid
  Arms: ENLDEPA
Drug: Placebo — The subjects take in 24 pils of gelatin capsule (each contains 0.25g of olive oil, provided by nutritional department of our institute) per day. The treatment lasts for 21d.
  Other Names: Gelatin capsule
  Arms: EN
Drug: HDEPA — The subjects take in 24 pils of EPA capsule per day. The medium is gelatine. Each capsule contains 0.25g of EPA. The capsules are provided by nutritional department of our institute). The treatment lasts for 21d.
  Other Names: Eicosapentaenoic acid
  Arms: ENHDPEA
Drug: Chemotherapy — Oxaliplatin 135mg/m2 d1，xeloda 1000mg/m2 d1-21. (XELOX)
  Other Names: XELOX chemotherapy

SUMMARY:
Malnutrition is frequently seen in patients on chemotherapy suffering from gastric/colorectal cancer and may worsen the outcome. EPA, a sort of ω-3 PUFA, can modulate immune system. EPA also antagonizes metabolic and inflammatory changes induced by the tumor. This study is to test whether EPA, in combination with enteral nutrition, can improve nutritional/immunologic status, quality of life, and reduce chemotherapy related side effects of these patients.

DETAILED DESCRIPTION:
Chemotherapy is indispensible for patients suffering from advanced gastric or colorectal cancer, and also the main therapy for those with end-stage tumor. However, incidence of malnutrition during chemotherapy was reported as high as 60%. The mechanisms include anatomy modification of digestive tract, side effects of chemotherapy such as anorexia, nausea, vomiting, and inflammatory factors generated or induced by the tumor. Malnutrition may lead to discontinuation of the therapy, compromise of the anti-cancer effect, increase of toxicity and mortality. 20%-40% of patients with end-stage tumor ultimately died from malnutrition.

EPA (Eicosapentaenoic acid, molecular formula C20H30O2) belongs to ω-3 polyunsaturated fatty acid (ω-3 PUFA). EPA is one of the main constituent of fish oil. EPA decreases LPS-stimulated macrophage production of TNF-α, IL-1β, IL-6, and human B lymphocytes production of IL-10, TNF-α, IFN-γ. EPA can suppress cancer induced lipolysis, and enhanced the inhibitory effect of 5-Fu over cancer cell proliferation. However, cancer patients are always lack of EPA.

Nutriall is a sort of non-elemental diet. The kind of powder is produced by Guangdong Academy of Agriculture Science. Every 50 grams of nutriall contains 9.3mg of VitC and 0.8mg of VitE. For this enteral nutrition preparation, there have been evidences of protective effects on nutritional status during chemotherapy on lung cancer. However, this kind of preparation does not contain EPA.

Up to date, there has been no RCT which testified whether therapeutic dosage of EPA plus enteral nutrition has combined effects on patients receiving chemotherapy. The investigators choose nutriall as basic nutritional support agent during chemotherapy, and give patients different dosage of EPA. Nutritional and immunologic status, quality of life and side effects of chemotherapy are recorded to evaluate whether EPA can improve outcome of these patients. Through this study the investigators may also optimize the dose of EPA for patients receiving chemotherapy on gastric/colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* The cases have undergone radical excision on gastric cancer or colorectal cancer.
* Without contraindication for chemotherapy.
* Eligible for postoperative adjuvant XELOX chemotherapy.
* Capable of taking in food or drug orally.
* Without severe absorption dysfunction
* Able and willing to give written, informed consent

Exclusion Criteria:

* Comorbidities: diseases of hematology or immunology system; hepatic or renal dysfunction; metabolic diseases.
* BMI>35kg/m2
* Life expectancy≤3mo
* The chemotherapy treatment is palliative.
* The patient has received radiotherapy or neoadjuvant chemotherapy prior to the operation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-12 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Serum level of proalbumin | The starting and ending day of the experiment for a certain subject (day1 and day21)

SECONDARY OUTCOMES:
Weight in light clothing | The starting and ending day of the experiment for a certain subject (day1 and day21)
Height and BMI | The starting and ending day of the experiment for a certain subject (day1 and day21)
mid upper arm circumference and triceps skinfold thickness | The starting and ending day of the experiment for a certain subject (day1 and day21)
Fat ratio and fat mass | The starting and ending day of the experiment for a certain subject (day1 and day21)
Fat-free mass, muscle mass and muscle function | The starting and ending day of the experiment for a certain subject (day1 and day21)
CD distribution of T cells | The starting and ending day of the experiment for a certain subject (day1 and day21)
Serum level of different types of immunoglobulin | The starting and ending day of the experiment for a certain subject (day1 and day21)
Serum level of different types of cytokines | The starting and ending day of the experiment for a certain subject (day1 and day21)
Serum level of Cortisol | The starting and ending day of the experiment for a certain subject (day1 and day21)
Serum level of transferrin | The starting and ending day of the experiment for a certain subject (day1 and day21)
Serum level of ALT and AST | The starting and ending day of the experiment for a certain subject (day1 and day21)
Serum level of creatine and BUN | The starting and ending day of the experiment for a certain subject (day1 and day21)
Serum level of total triglyceride, total cholesterol, LDL, HDL | The starting and ending day of the experiment for a certain subject (day1 and day21)
Records of EPA intake | The whole experiment period
Records of chemotherapy-associated side effects | The whole experiment period
Serum level of albumin | The starting and ending day of the experiment for a certain subject (day1 and day21)
Serum level of CEA, CA125, CA199 | The starting and ending day of the experiment for a certain subject (day1 and day21)
Records of Nutriall intake | The whole experiment period
Records of food intake | The middle 3 days of the whole experiment period (day10, day11, day12)

CONTACTS AND LOCATIONS:
Overall Officials: Huilian Zhu, MD, Study Director — Sun Yat-sen University
Locations (1):
- First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Barber MD, Fearon KC. Tolerance and incorporation of a high-dose eicosapentaenoic acid diester emulsion by patients with pancreatic cancer cachexia. Lipids. 2001 Apr;36(4):347-51. doi: 10.1007/s11745-001-0726-4. PMID 11383684
- [Background] Bayram I, Erbey F, Celik N, Nelson JL, Tanyeli A. The use of a protein and energy dense eicosapentaenoic acid containing supplement for malignancy-related weight loss in children. Pediatr Blood Cancer. 2009 May;52(5):571-4. doi: 10.1002/pbc.21852. PMID 19090549
- [Background] Calviello G, Di Nicuolo F, Serini S, Piccioni E, Boninsegna A, Maggiano N, Ranelletti FO, Palozza P. Docosahexaenoic acid enhances the susceptibility of human colorectal cancer cells to 5-fluorouracil. Cancer Chemother Pharmacol. 2005 Jan;55(1):12-20. doi: 10.1007/s00280-004-0846-6. Epub 2004 Sep 10. PMID 15365767
- [Background] Crooks V, Waller S, Smith T, Hahn TJ. The use of the Karnofsky Performance Scale in determining outcomes and risk in geriatric outpatients. J Gerontol. 1991 Jul;46(4):M139-44. doi: 10.1093/geronj/46.4.m139. PMID 2071835
- [Background] Elia M, Van Bokhorst-de van der Schueren MA, Garvey J, Goedhart A, Lundholm K, Nitenberg G, Stratton RJ. Enteral (oral or tube administration) nutritional support and eicosapentaenoic acid in patients with cancer: a systematic review. Int J Oncol. 2006 Jan;28(1):5-23. doi: 10.3892/ijo.28.1.5. PMID 16327975
- [Background] Gorjao R, Azevedo-Martins AK, Rodrigues HG, Abdulkader F, Arcisio-Miranda M, Procopio J, Curi R. Comparative effects of DHA and EPA on cell function. Pharmacol Ther. 2009 Apr;122(1):56-64. doi: 10.1016/j.pharmthera.2009.01.004. Epub 2009 Feb 12. PMID 19318040
- [Background] Pratt VC, Watanabe S, Bruera E, Mackey J, Clandinin MT, Baracos VE, Field CJ. Plasma and neutrophil fatty acid composition in advanced cancer patients and response to fish oil supplementation. Br J Cancer. 2002 Dec 2;87(12):1370-8. doi: 10.1038/sj.bjc.6600659. PMID 12454764
- [Background] Read JA, Beale PJ, Volker DH, Smith N, Childs A, Clarke SJ. Nutrition intervention using an eicosapentaenoic acid (EPA)-containing supplement in patients with advanced colorectal cancer. Effects on nutritional and inflammatory status: a phase II trial. Support Care Cancer. 2007 Mar;15(3):301-7. doi: 10.1007/s00520-006-0153-3. Epub 2006 Oct 5. PMID 17021855
- [Background] Read JA, Crockett N, Volker DH, MacLennan P, Choy ST, Beale P, Clarke SJ. Nutritional assessment in cancer: comparing the Mini-Nutritional Assessment (MNA) with the scored Patient-Generated Subjective Global Assessment (PGSGA). Nutr Cancer. 2005;53(1):51-6. doi: 10.1207/s15327914nc5301_6. PMID 16351506
- [Background] Russell ST, Tisdale MJ. Effect of eicosapentaenoic acid (EPA) on expression of a lipid mobilizing factor in adipose tissue in cancer cachexia. Prostaglandins Leukot Essent Fatty Acids. 2005 Jun;72(6):409-14. doi: 10.1016/j.plefa.2005.03.002. PMID 15899583
- [Background] Wang ZD, Peng JS, Chen S, Huang ZM, Huang L. [Effects of perioperative enteral immunonutrition on nutritional status, immunity and inflammatory response of elderly patients]. Zhonghua Yi Xue Za Zhi. 2006 May 30;86(20):1410-3. Chinese. PMID 16796925
- [Background] Yam D, Peled A, Shinitzky M. Suppression of tumor growth and metastasis by dietary fish oil combined with vitamins E and C and cisplatin. Cancer Chemother Pharmacol. 2001;47(1):34-40. doi: 10.1007/s002800000205. PMID 11221959
- [Background] Zhong HJ, Ying JE, Ma SL. [Effect of Supportan on nutritional status and immune function of late-staged gastric cancer patients undergoing chemotherapy]. Zhonghua Wei Chang Wai Ke Za Zhi. 2006 Sep;9(5):405-8. Chinese. PMID 17043961